CLINICAL TRIAL: NCT03703622
Title: The Effect of Standard Helping Babies Breathe Training With Video-debriefing on Health Workers Knowledge and Skills Attainment and Retention in Lira District Northern Uganda
Brief Title: Video-Debriefing for Improved Competence Among Skilled Birth Attendants in Lira District-Northern Uganda
Acronym: V-DICAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: REC REF 2015-085
Record Dates: First submitted 2018-09-28; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Neonatal Encephalopathy; Helping Babies Breathe (HBB) Training
Keywords: HBB knowledge and skills attainment and retention; Video-debriefing; Skills, knowledge, Birth attendants

STUDY DESIGN:
Intervention Model Description: The AAP HBB curriculum will be used to train participants. Lectures will be delivered by the PI (Master Trainers), followed by demonstration of HBB skills using NeoNatali Mannequin. The participants will then be divided into two groups. One group for practical sessions with master trainers and the other group video-debriefing. The video-debriefing group will have their practical sessions filmed and then the film used for debriefing feedback. First the experiences of the team performing resuscitation will be obtained then positive feedback and learning points from other learners will be given in a respectful safe environment. All participants will be encouraged to contribute in the discussion. Pre- and Post-Test knowledge and skills will be assessed will be done using MCQs, and bag mask ventilation, OSCE A and B checklists from 2nd edition AAP HBB training manual.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cluster randomization was done by an independent statistician from the University of Bergen who is not part of the study. The health workers from randomised facilities were randomly assigned to two groups of 24 participants, each to be trained for two days. The participants and the assessors did not know the intervention groups which they belonged to until the day of training. During follow-up the assessors and the PI will not know which intervention arms the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-debriefing with standard HBB training (Experimental): Health workers are given standard HBB training according to American Association of Pediatrics (AAP) plus video-debriefing. Filming of the simulated case scenarios will be done and after which the films will be used for debriefing or feedback. Participants will be encouraged to give feedback with the guidance of master trainer and the PI. Teams of three participants(birth attendant, mother and helper) will perform the HBB simulation or scenarios. After each scenario, debriefing is done until all participants have had the opportunity to participate in the simulation exercise. All the participants in this arm will undergo HBB practical sessions such as bag mask ventilation skills sessions, care of the health new-born and sick newborn baby who needs resuscitation care. Pre and post-tests will be done to assess performance of all participants.
  Interventions: Behavioral: Video-debriefing with standard HBB training compared with standard HBB training only
- Standard HBB training only (Active Comparator): Health workers are given standard HBB training according to AAP without video-debriefing. All the participants in this arm, like in intervention arm, will also undergo HBB practical sessions such as bag mask ventilation skills sessions, care of the health new-born and sick new-born baby who needs resuscitation care only. Pre-and post-tests will be done to assess performance of all participants.
  Interventions: Behavioral: Video-debriefing with standard HBB training compared with standard HBB training only

INTERVENTIONS:
Behavioral: Video-debriefing with standard HBB training compared with standard HBB training only — We will use the AAP training curriculum for the HBB 2nd edition through out the training and course assessments pre-and post- training and during follow-up period.
  Both intervention arms will a 2 days training consisting of: lectures, neonatal resuscitation demonstrations using NeoNatali mannequin, and practical skills s sessions. Pre- and post-tests knowledge (MCQs) and skills (bag mask ventilation, OSCE A, & OSCE B) will be given to all participants.
  In the intervention arm, in addition to standard training, participants will work in teams of three (birth attendant, mother, and an assistant) to perform different HBB case scenarios. These will be filmed and used for subsequent debriefing after each case scenarios. After all participants in the intervention have had the opportunity to participate in the debriefing, then a post test is done to assess performance.
  Analysis is done to compare the intervention and control arms performances.

SUMMARY:
Helping babies breathe (HBB) is a neonatal resuscitation training program for low-resource settings to health care workers to provide prompt respiratory support to save babies at birth. Despite massive roll-out, new-born mortality reduction has stagnated over the years. Innovative teaching methods with existing technology such as video-debriefing needs to be tested to promote competence (skills and knowledge) attainment and retention.

DETAILED DESCRIPTION:
In this study we will randomize both public and private delivery facilities in Lira district northern Uganda to receive either standard HBB with video-debriefing (intervention) or standard training alone (control). We hope video-debriefing will improve competence among the health workers and promote skills and knowledge retention over time, hence reduction in neonatal mortality.

The result of the study may also contribute to shaping refresher training program policy in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* All health care workers attending to delivery and new-born care in both public and private facilities in Lira district.

Exclusion Criteria:

* Those who turn up for training just for daily allowances, having been sent by their facility in-charges to fill gaps such as community vaccinators, Village Health Teams (VHTs), security officers, cleaners, and laboratory technicians

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Health workers knowledge scores in percentage | 6 months
  The scores from HBB multiple choice questions (MCQs) will be used.
Health workers skills scores in percentages | 6 months
  The scores from bag mask ventilation, OSCE A and B skills sessions will be used.

SECONDARY OUTCOMES:
Knowledge and skills retention at 1, 3 and 6 months | 6 months
  The knowledge and skills scores as described above will be used to assess retention at different time points
Neonatal mortality at health facilities pre- and post training | 6 months
  We will determine the mortality at all the birth facilities from maternity registers to determine the effect of our training on birth outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- All public and Private delivery facilities (hospitals, health centers, maternity homes, and clinics) in Lira district, Lira, Northern Region, Uganda

IPD SHARING:
Plan to Share IPD: Yes
After dissemination and Doctor of Philosophy (PhD) defence, I can avail the scores and demographics of the study participants after de-identification of the dataset.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 months
Access Criteria: Direct contact to the PI

REFERENCES:
- [Derived] Odongkara B, Tylleskar T, Pejovic N, Achora V, Mukunya D, Ndeezi G, Tumwine JK, Nankabirwa V. Adding video-debriefing to Helping-Babies-Breathe training enhanced retention of neonatal resuscitation knowledge and skills among health workers in Uganda: a cluster randomized trial. Glob Health Action. 2020 Dec 31;13(1):1743496. doi: 10.1080/16549716.2020.1743496. PMID 32524895